CLINICAL TRIAL: NCT00242268
Title: A Safety Study of Combination Treatment With Avonex and Zocor in Relapsing Remitting Multiple Sclerosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alabama Neurology Associates, PC (Other)
Collaborators: Biogen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IST 03-09
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2005-12-07 (Estimated); Status verified 2005-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
The purpose of this study is to determine if using Avonex in combination with Zocor is a safe and effective therapy for subjects with relapsing remitting multiple sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an inflammatory demyelinating disease of the Central Nervous System (CNS). There are many forms of MS; althoughthe majority are Relapsing Remitting (RRMS) representing approximately 80% of the cases. The disease appears to be more inflammatory in RRMS as manisfested by an increase inGadolinium enhancement on MRI and an increase in inflammatory bioassay markers.

Zocor is in a class of drugs (statins) that are used to lower cholesterol. Statins also have an anti-inflammatory effect on the CNS. Zocor has been shown in a small clinical trial to reduce the number of new MRI-detected brain lesions over a six month treatment period in patients with RRMS. This study is to evaluate the safety of combining Avonex with Zocor for a a period of fourteen months in patients with RRMS and to evaluate the effect of treatment on new or enlarging lesions as measured by MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant females age 18-55 who have clinically and laboratory definite relapsing-remitting MS using the MacDonald criteria.
2. Subjects must be taking some form of interferon therapy (Rebif, Avonex or Betaseron) for a duration of 12 months with documented breakthrough disease as defined:

   * or = 1 documented clinical relapse in past 12 months while on interferon therapy. For eligibility, a pre-study relapse is defined as neurologic symptoms and signs documented by review of the history with the subject or in the medical record, of sufficient severity and duration to be determined by the investigator as consistent with an acute MS relapse.

   The relapse does not need to have been treated to qualify. the timing of the relapse is defined based on the onset of symptoms.

   OR

   > or = 1 documented Gd-enhancing lesion on cranial or spinal MRI. The presence of a Gd-enhancing lesion must be documented either by a report in the medical record or review of the films by the investigator.
3. The Kurtzke EDSS score must be between 0- 5.0.
4. All subjects must give written consent prior to evaluation and testing.

Exclusion Criteria:

1. Subjects with primary or secondary progressive MS.
2. Female patients may not be pregnant, attempting pregnancy or breastfeeding.
3. Female subjects must use an acceptable form of contraception during the study as defined by the investigators. The rhythm method is not to be used as the sole method of contraception.
4. Subjects unwilling or unable to give informed consent.
5. Subjects that are NAB+ (titers > or = 20).
6. Abnormal baseline blood test exceeding any of the limits defined below:

   1. ALT or AST > 2x upper limit of normal (ULN)
   2. CPK > 2x upper limit of normal (ULN)
   3. Total WBC < 3,000/mm3
7. No chronic infections (including HIV and Hepatitis B/C) may be present.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-10

PRIMARY OUTCOMES:
1. To evaluate the safety of combining Avonex with Zocor for a period of fourteen months in patients with RRMS
2. To evaluate the effect of treatment on MRI, specifically new or enlarging T2 lesions burden

SECONDARY OUTCOMES:
1. To evaluate the effect on Relapse Rates
2. To evaluate the effect on disease progression as measured with EDSS and MSFC

CONTACTS AND LOCATIONS:
Overall Officials: Emily S. Riser, MD, Principal Investigator
Locations (1):
- Alabama Neurology Associates, Birmingham, Alabama, United States